CLINICAL TRIAL: NCT07286344
Title: Effect of Fluoride Varnish Formulation on the Management of Dentin Hypersensitivity: A Randomized Clinical Trial
Brief Title: Effect of Fluoride Varnish Formulation on the Management of Dentin Hypersensitivity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Concepcion, Chile (Other)
Collaborators: Solventum (Industry)
Responsible Party: Principal Investigator, Michael Wendler Ernst, Associate Professor, University of Concepcion, Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEC-SSC 25-10-120
Record Dates: First submitted 2025-12-10; First posted 2025-12-16 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Hypersensitivity Dentin; Fluoride Varnishes
Keywords: Dentin hypersensitivity; Fluoride varnishes; Visual analogue scale (VAS); Schiff scale; OHIP-14; Desensitizing agents; Aqueous fluoride varnish
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial with parallel arms
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Resin/rosin-based varnish, 22,600 ppm NaF (Duraphat® Fluoride Varnish) (Active Comparator): Application procedure:
  * The tooth surface will be cleaned and saliva gently removed.
  * The appropriate amount of varnish will be dispensed onto an application tray.
  * The varnish will be applied with a cotton applicator, probe, or brush, forming a thin film.
  * The patient will remain seated with lip retractors in place for 15 minutes.
  * Patients will be instructed not to brush their teeth or chew hard foods for at least 4 hours post-application.
  Interventions: Device: Resin/rosin-based varnish, 22,600 ppm NaF
- Aqueous fluoride varnish, 9,500 ppm NaF (Clinpro Clear® Fluoride Varnish) (Experimental): Application procedure:
  * The tooth surface will be cleaned and dried; a lip retractor will be used.
  * The varnish will be expressed fully into the dispensing chamber of the unit-dose package.
  * Using the applicator brush, the varnish will be applied to fully cover the hypersensitive area.
  * Patients will be instructed not to touch the teeth with the tongue or attempt to remove the varnish.
  * After application, patients will remain with lip retractors in place for 15 minutes.
  Interventions: Device: Aqueous fluoride varnish, 9,500 ppm NaF

INTERVENTIONS:
Device: Aqueous fluoride varnish, 9,500 ppm NaF — The tooth surface will be cleaned and dried with a lip retractor in place. The varnish will be dispensed into the unit-dose chamber and applied with a brush to fully cover the hypersensitive area. Patients will be instructed not to disturb the varnish and will remain with the lip retractors in place for 15 minutes.
  Arms: Aqueous fluoride varnish, 9,500 ppm NaF (Clinpro Clear® Fluoride Varnish)
Device: Resin/rosin-based varnish, 22,600 ppm NaF — The tooth surface will be cleaned and dried, and the varnish will be dispensed onto an application tray. A thin film will be applied using a cotton applicator, probe, or brush. Patients will remain seated with lip retractors in place for 15 minutes and will be advised to avoid toothbrushing and hard foods for at least 4 hours after application.
  Arms: Resin/rosin-based varnish, 22,600 ppm NaF (Duraphat® Fluoride Varnish)

SUMMARY:
This randomized controlled clinical trial aims to determine whether different fluoride varnish formulations reduce dentin hypersensitivity (DH) in young adults diagnosed with DH. The primary purpose of this study is to evaluate the clinical effectiveness of two commercially available fluoride varnishes.

The main questions this study aims to answer are:

* Does Clinpro Clear® (aqueous base, 9,500 ppm NaF) lead to a greater reduction in dentin hypersensitivity compared with Duraphat® (rosin/resin base, 22,600 ppm NaF)?
* Do these varnish formulations improve oral health-related quality of life and patient satisfaction?

Researchers will compare a single application of Duraphat® with a single application of Clinpro Clear® to assess differences in hypersensitivity reduction, quality-of-life outcomes, and patient satisfaction.

Participants will:

* Receive one application of either Duraphat® or Clinpro Clear® under standardized clinical conditions.
* Complete baseline and post-treatment evaluations, including:
* Dentin hypersensitivity intensity using a visual analogue scale (VAS)
* Air-blast response using the Schiff scale
* Oral health-related quality of life using the OHIP-14
* Patient satisfaction using the CSAT survey

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40 years
* Absence of systemic diseases with oral manifestations or requiring medications with antisialagogue effects
* Fully dentate (excluding third molars or teeth extracted for orthodontic reasons)
* Absence of periodontal disease, or periodontal condition in a stable state
* Presence of at least one cervical lesion with a Schiff sensitivity score ≥ 1
* No previous treatment or restorative procedures on the target lesions (including no topical fluoride application within the last 6 months)

Exclusion Criteria:

* Patients requiring long-term use of NSAIDs or other analgesic/anti-inflammatory medications
* Patients with allergy to milk proteins
* Patients with allergy to organic resins or pine-derived substances
* Pregnant or breastfeeding individuals
* Patients with fixed orthodontic appliances in place

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2026-05-29 (Estimated); Study Completion 2026-06-26 (Estimated)

PRIMARY OUTCOMES:
Change in dentin hypersensitivity to mechanical stimulation from baseline to post-fluoride varnish application | Baseline; 7 and 28 days after the intervention.
  Visual Analogue Scale (VAS) With the tooth isolated and dry, a curved dental probe will be gently passed in a mesiodistal direction across the lesion area. Pain perception will be assessed using a VAS, on which the patient indicates the perceived pain intensity, ranging from no pain (0) to the worst pain imaginable (100). The score, measured on a 0-100 mm scale, will be recorded for each lesion.
Change in dentin hypersensitivity to air stimulation from baseline to post-fluoride varnish application | Baseline; 7 and 28 days after the intervention.
  Air blast test (Schiff test)
  An air stimulus will be applied for 4 seconds from a distance of 3-4 mm using a triple syringe with standardized air pressure (40-60 psi) at room temperature. In cases of cervical lesions on adjacent teeth, neighboring lesions will be isolated with cotton to ensure tooth-specific responses. Pain response will be assessed using the Schiff sensitivity scale:
  * Score 0: No response to the air stimulus.
  * Score 1: A response is perceived, but the subject does not request discontinuation of the stimulus and does not move away.
  * Score 2: A response is perceived and the subject requests discontinuation of the stimulus or involuntarily moves away.
  * Score 3: An intense pain response occurs, with immediate request to stop the stimulus or marked withdrawal from it.

SECONDARY OUTCOMES:
Change in oral health-related quality of life from baseline to post-fluoride varnish application | Baseline; 28 days after intervention
  This outcome will be measured using a validated translation to Spanish of the Oral Health Impact Profile (OHIP-14), evaluating the impact of dentin hypersensitivity on quality of life across seven domains: functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability, and handicap. Patients report how frequently they experienced dentin hypersensitivity-related problems using a 5-point Likert scale (0 = never to 4 = very often). Total scores range from 0-56, with higher scores indicating poorer oral health-related quality of life.
Patient satisfaction following fluoride varnish application | 7 days after intervention.
  Client Satisfaction Assessment Tool (CSAT) CSAT will assess patient satisfaction using three items evaluating comfort during fluoride varnish application, ease of adherence to post-application instructions, and likelihood of recommending the treatment to others with dentin hypersensitivity. Each item is rated on a 5-point Likert scale ranging from negative to positive perceptions (1 = very uncomfortable/difficult/improbable to 5 = very comfortable/easy/probable), with higher scores indicating greater patient satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Muñoz, DDS, Principal Investigator — Department of Restorative Dentistry, Faculty of Dentistry, Universidad de Concepcion; Michael Wendler, DDS, PhD, Study Director — Department of Restorative Dentistry, Faculty of Dentistry, Universidad de Concepcion
Locations (1):
- Clinica de Rehabilitación Avanzada e Implantologia (CRAI), Concepción, Región del Biobío, Chile

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. Only aggregated and de-identified summary data may be included in publications and scientific presentations. IPD will not be shared because the study is small in scale, involves sensitive clinical information, and sharing participant-level data may pose privacy risks that cannot be fully mitigated. Additionally, the research objectives can be addressed through summary-level reporting without requiring access to individual datasets.

REFERENCES:
- [Result] Tenuta LMA, Capalbo LC, Yoshino EY. Enamel Fluoride Reactivity of Professional Fluoride Products Is Not Correlated With Their Total Fluoride Content. Pediatr Dent. 2025 May 15;47(3):178-182. PMID 40533917
- [Result] Sharan A, Pawar B, Bagde H, Chawla TK, Dhan AV, Shyamsukha B, Sharma S. Comparative Evaluation of Dentin Hypersensitivity Reduction Over One Month after a Single Topical Application of Three Different Materials: A Prospective Experimental Study. J Pharm Bioallied Sci. 2024 Dec;16(Suppl 4):S3405-S3407. doi: 10.4103/jpbs.jpbs_848_24. Epub 2024 Oct 29. PMID 39926954
- [Result] Sgreccia PC, Dame-Teixeira N, Barbosa RES, Araujo PF, Zanatta RF, Garcia FCP. Assessment of the Oral Health Impact Profile (OHIP-14) improvement of different treatments for dentin hypersensitivity in noncarious cervical lesions-a randomized clinical study. Clin Oral Investig. 2022 Nov;26(11):6583-6591. doi: 10.1007/s00784-022-04610-x. Epub 2022 Jul 7. PMID 35796800
- [Result] Porto IC, Andrade AK, Montes MA. Diagnosis and treatment of dentinal hypersensitivity. J Oral Sci. 2009 Sep;51(3):323-32. doi: 10.2334/josnusd.51.323. PMID 19776498
- [Result] Machado AC, Maximiano V, Yoshida ML, Freitas JG, Mendes FM, Aranha ACC, Scaramucci T. Efficacy of a calcium-phosphate/fluoride varnish and ionomeric sealant on cervical dentin hypersensitivity: A randomized, double-blind, placebo-controlled clinical study. J Oral Rehabil. 2022 Jan;49(1):62-70. doi: 10.1111/joor.13270. Epub 2021 Nov 2. PMID 34676918
- [Result] Lopez R, Baelum V. Spanish version of the Oral Health Impact Profile (OHIP-Sp). BMC Oral Health. 2006 Jul 7;6:11. doi: 10.1186/1472-6831-6-11. PMID 16827940
- [Result] Garofalo SA, Sakae LO, Machado AC, Cunha SR, Zezell DM, Scaramucci T, Aranha AC. In Vitro Effect of Innovative Desensitizing Agents on Dentin Tubule Occlusion and Erosive Wear. Oper Dent. 2019 Mar/Apr;44(2):168-177. doi: 10.2341/17-284-L. Epub 2018 Jun 28. PMID 29953338
- [Result] Fernandez CE, Tenuta LM, Zarate P, Cury JA. Insoluble NaF in Duraphat(R) may prolong fluoride reactivity of varnish retained on dental surfaces. Braz Dent J. 2014;25(2):160-4. doi: 10.1590/0103-6440201302405. PMID 25140722
- [Result] Douglas-de-Oliveira DW, Vitor GP, Silveira JO, Martins CC, Costa FO, Cota LOM. Effect of dentin hypersensitivity treatment on oral health related quality of life - A systematic review and meta-analysis. J Dent. 2018 Apr;71:1-8. doi: 10.1016/j.jdent.2017.12.007. Epub 2017 Dec 17. PMID 29262305
- [Result] Dall Agnol MA, Battiston C, Tenuta LMA, Cury JA. Fluoride Formed on Enamel by Fluoride Varnish or Gel Application: A Randomized Controlled Clinical Trial. Caries Res. 2022;56(1):73-80. doi: 10.1159/000521454. Epub 2021 Dec 13. PMID 34915485